CLINICAL TRIAL: NCT03005665
Title: Effect of Orogastric Acetazolamide on Intraocular Pressure in Laparoscopic Donor Nephrectomies
Brief Title: Effect of Acetazolamide on Optic Nerve Sheath Diameter in Laparoscopic Donor Nephrectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Ashish Singh Aditya, JUNIOR RESIDENT, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10055/PG-2Trg/2014/24258-59
Record Dates: First submitted 2016-12-15; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Intracranial Pressure Increase
Keywords: optic nerve sheath diameter; acetazolamide
MeSH Terms: conditions — Intracranial Hypertension | interventions — Acetazolamide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Acetazolamide (Experimental): Acetazolamide 5 mg/kg diluted in 10 ml normal saline through orogastric Ryle's Tube soon after the induction of anaesthesia followed by 10 ml normal saline flush.
  Interventions: Drug: Acetazolamide
- Group s - Normal saline (Placebo Comparator): 20 ml normal saline total volume.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Group A - Acetazolamide
Drug: Normal Saline
  Arms: Group s - Normal saline

SUMMARY:
The purpose of the trial is to study the effect of acetazolamide administered via Ryle's tube on optic nerve sheath diameter in laparoscopic live donor nephrectomy patients.

DETAILED DESCRIPTION:
this study was done on 40 American Society of Anaesthesiologist(ASA) I & II live donors of either sex in adult age group undergoing laparoscopic live donor nephrectomy. After getting approval from institutes ethical committee and written informed consent, Donors were randomly allocated to either of two group. Anaesthesia was induced with injection morphine 0.1 mg/kg, injection propofol 1-2 mg/kg and vecuronium 0.1 mg/kg. Maintenance of anaesthesia was done with isoflurane and oxygen. After induction donors were placed into modified flank position with left side upward. Donors in Group A received Acetazolamide 5 mg/kg via orogastric tube soon after the induction of anaesthesia. Group S received saline as a placebo. investigator and subjects were blinded till the statistical analysis. Optic nerve sheath diameter was measured six times during perioperative periods by using high frequency ultrasound probe. Intra operative monitoring was done for Heart rate, Blood Pressure, pulse oximetry(Spo2), End Tidal Carbon Dioxide(ETCO2), Train Of Four(TOF) and Bi spectral index(BIS). Post operatively donors were reversed with injection neostigmine and glycopyrrolate.

once return of spontaneous ventilation was well established and patient becomes conscious oriented trachea was extubated and donors were shifted to post anaesthetic care unit(PACU). Postoperatively donors were monitored for Heart rate, Blood Pressure, Spo2, Comfort Score, Visual analog score for incisional site pain and shoulder tip pain, and Post operative nausea vomiting. Rescue analgesia was given to patients having comfort score less than 6.

After completion of study Optic nerve sheath diameter, pain scores and comfort scores was compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* 18-60 years of age
* Hemodynamically stable patients.

Exclusion Criteria:

* Patient's refusal.
* Ocular Defects/ Wounds /Previous ocular surgery.
* H/O Hypertension
* Patients having Double Renal Arteries.
* Laparoscopic Nephrectomies converted to Open Surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Optic nerve sheath diameter being assessed | baseline, 5 minutes, 10 minutes, 60 minutes, 120 minutes, 5 minutes post surgery
  optic nerve sheath diameter measured during perioperative period

SECONDARY OUTCOMES:
Visual analog score for incision site and shoulder pain | baseline, 30 minutes, 60 minutes, 4 Hours, 12 hours, 24 Hours, 48 hours, 72 Hours.
  visual analog score will be monitored postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ashish S Aditya, MD, Principal Investigator — PGIMER, chandigarh, INDIA
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India